CLINICAL TRIAL: NCT04997629
Title: Preserve Biological Samples and Gene Extracts of All Sports Medicine-related Diseases. To Study Related Gene Mutation Sites and Regulation. To Study Related Molecular Mechanisms and Signaling Pathways. A Storage Platform for Sports Medicine-related Diseases Research Sample Database Has Been Established.
Brief Title: Gene Biobank of Sports Injuries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2019063
Record Dates: First submitted 2021-06-27; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-06

CONDITIONS: Gene Insertions; Gene Deletion
Keywords: sports medicine; platform; sample database; gene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preserve biological samples and gene extracts of all sports medicine-related diseases. To study related gene mutation sites and regulation. To study related molecular mechanisms and signaling pathways. A storage platform for sports medicine-related diseases research sample database has been established.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with joint sports injuries.
2. Follow-up patients after sports injury.
3. Patients with genetic predisposition to sports injuries.
4. Patients with family genetic predisposition to exercise-related diseases and their relatives.

Exclusion Criteria:

1. Patients with joint damage caused by external force.
2. The patient is accompanied by other injuries at the same time.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients related to sports injuries
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Magnetic resonance imaging (MRI) | Before the operation
  All MRI scans were obtained with a 3.0-T MRI scanner (Magnetom Trio with TIM system, Siemens Healthcare). Five routine MRI sequences with a section thickness of 4 mm were obtained in all patients. Preoperative and postoperative evaluations of the articular cartilage of the transplanted compartment were performed with the Yulish score41 (grade 0 = normal; grade 1 = normal contour 6 abnormal signal; grade 2 = superficial fraying, erosion, or ulceration of <50%; grade 3 = partial-thickness defect of >50% but <100%; grade 4 = full-thickness cartilage loss). The signal of the meniscus allograft in the coronal plane of the T2-weighted fast spin echo sequence was graded on a scale of 0 to 3.
Magnetic resonance imaging (MRI) | an average of 1 year
  All MRI scans were obtained with a 3.0-T MRI scanner (Magnetom Trio with TIM system, Siemens Healthcare). Five routine MRI sequences with a section thickness of 4 mm were obtained in all patients. Preoperative and postoperative evaluations of the articular cartilage of the transplanted compartment were performed with the Yulish score41 (grade 0 = normal; grade 1 = normal contour 6 abnormal signal; grade 2 = superficial fraying, erosion, or ulceration of <50%; grade 3 = partial-thickness defect of >50% but <100%; grade 4 = full-thickness cartilage loss). The signal of the meniscus allograft in the coronal plane of the T2-weighted fast spin echo sequence was graded on a scale of 0 to 3.
Radiographs | Before the operation
  All patients also obtained 45° flexion weightbearing AP radiographs of both the ipsilateral and contralateral sides at final follow-up. The radiograph of the total length of the lower limbs was used to evaluate alignment. In the AP plain radiographs, the shortest distance between the femoral condyle and tibial plateau of the transplanted side was measured and designated as the joint space height. The difference between the ipsilateral and contralateral sides was calculated to identify joint space narrowing. In addition, Kellgren-Lawrence (K-L) grading was used to assess the osteoarthritic status of the knee.
Radiographs | an average of 1 year
  All patients also obtained 45° flexion weightbearing AP radiographs of both the ipsilateral and contralateral sides at final follow-up. The radiograph of the total length of the lower limbs was used to evaluate alignment. In the AP plain radiographs, the shortest distance between the femoral condyle and tibial plateau of the transplanted side was measured and designated as the joint space height. The difference between the ipsilateral and contralateral sides was calculated to identify joint space narrowing. In addition, Kellgren-Lawrence (K-L) grading was used to assess the osteoarthritic status of the knee.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Lin, Study Director — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China